CLINICAL TRIAL: NCT05130281
Title: Mobile Cognitive Behavior Therapy Targeting Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1803019086
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Anxiety Disorders and Symptoms
Keywords: anxiety; mental health; adolescents; young adults; CBT; mobile app; Cognitive Behavior Therapy
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial designed to assess the feasibility of Maya, an app-based CBT intervention, and provide preliminary efficacy data for three different incentive strategies. Participants will be randomized to one of three incentive conditions: 1) a social support condition, 2) a gain-framed condition in which participants can earn "points" for completing assigned therapy sessions, and 3) a loss-framed condition in which participants begin with a specified number of points that they can lose for failing to complete assigned therapy sessions on time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Support (Experimental): Participants receive treatment with the Maya app in conjunction with social support incentives for 6 weeks.
  Interventions: Behavioral: Maya mobile app; Behavioral: Social Support
- Gain Framed (Experimental): Participants receive treatment with the Maya app in conjunction with gain-framed incentives for 6 weeks.
  Interventions: Behavioral: Maya mobile app; Behavioral: Gain Framed
- Loss Framed (Experimental): Participants receive treatment with the Maya app in conjunction with loss-framed incentives for 6 weeks.
  Interventions: Behavioral: Maya mobile app; Behavioral: Loss Framed

INTERVENTIONS:
Behavioral: Maya mobile app — The Maya app teaches cognitive behavioral therapy (CBT) techniques including emotion monitoring, cognitive restructuring, mindfulness, and exposure to help individuals with anxiety.
Behavioral: Social Support — Participants earn points and badges for completing sessions, homework, and skills on time and receive post session feedback via text message. Participants can identify a person they know to receive updates about their progress and support them throughout their time in the program. Participants will not be required to choose a person they know to receive updates about their use of the program; instead, they can choose to have a member of the study team serve as their social support if they are assigned to this condition.
  Arms: Social Support
Behavioral: Gain Framed — Participants earn points and badges for completing sessions, homework, and skills on time and receive post session feedback via text message.
  Arms: Gain Framed
Behavioral: Loss Framed — Participants lost points and badges for not completing sessions, homework, and skills on time and receive post session feedback via text message.
  Arms: Loss Framed

SUMMARY:
This study aims to examine different ways of motivating people to make use of Maya, a mobile cognitive behavior therapy (CBT) program for adolescents and young adults experiencing anxiety symptoms, and to assess whether social supports are as efficacious, or more efficacious, than other non-monetary incentives. Subjects will use the Maya app for at least 20 minutes per day, 2 days per week, for 6 weeks. Assessments will include a weekly check in with a member of the research team, questionnaires, and an optional magnetic resonance imaging (MRI) recording.

DETAILED DESCRIPTION:
There is a growing need for easily accessed anxiety treatments designed for young adults. Mobile app-based interventions can be disseminated more broadly than traditional psychosocial interventions and may be particularly appealing to this age group, which uses mobile devices frequently. Mobile apps can also collect real-time data about patient symptom severity and provide tailored, in-the-moment coping strategies.

This study aims to examine different ways of motivating people to make use of Maya, a mobile cognitive behavior therapy (CBT) app for adolescents and young adults experiencing anxiety symptoms, and to assess whether social supports are as efficacious, or more efficacious, than other non-monetary incentives. Young adults with anxiety will be randomized to one of three conditions: a social support condition, a gain-framed condition in which participants can earn "points" for completing their assigned sessions, and a loss-framed condition in which participants lose "points" for failing to complete their assigned sessions. Subjects will use the Maya app for at least 20 minutes per day, 2 days per week, for 6 weeks and will complete assessments at baseline, week 3, week 6 (end of treatment), and a follow-up assessment at week 12. Subjects may also choose to complete an optional magnetic resonance imaging (MRI) recording at the baseline and end of treatment (week 6).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 25
* Primary diagnosis of an anxiety disorder, as determined by a score of 4 on the Clinical Severity Rating from the Anxiety Disorders Interview Schedule (ADIS)

Exclusion Criteria:

* Score of < 4 on the ADIS
* Primary psychiatric diagnosis other than an anxiety disorder
* Currently in cognitive behavioral therapy outside of the study
* Change in dose of a psychiatric medication in the past 12 weeks
* Intent or plan to attempt suicide

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Gunning, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bress JN, Falk A, Schier MM, Jaywant A, Moroney E, Dargis M, Bennett SM, Scult MA, Volpp KG, Asch DA, Balachandran M, Perlis RH, Lee FS, Gunning FM. Efficacy of a Mobile App-Based Intervention for Young Adults With Anxiety Disorders: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2428372. doi: 10.1001/jamanetworkopen.2024.28372. PMID 39163044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through online advertisements, local college and university e-mail lists, and physical flyers posted across local colleges and universities between June 2021 and September 2022. The first particpant was enrolled 6/18/2021 and the last participant was enrolled 9/8/2022.
Pre-assignment Details: Eligible participants had a primary diagnosis of an anxiety disorder, were ages 18-25, and fluent in English. Exclusion criteria included current cognitive behavioral therapy, change in psychotropic medication dose in the past 12 weeks, or suicidal ideation with intent and/or plan. Of 68 people evaluated, 59 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Social Support | Gain Framed | Loss Framed
Started | 18 | 30 | 11
Completed | 18 | 30 | 10
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Support | Gain Framed | Loss Framed | Total
Number analyzed (Participants) | 18 | 30 | 11 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (1.2) | 22.9 (1.9) | 22.4 (2.4) | 23.1 (1.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 18 | 23 | 5 | 46
  Gender: Male | 0 | 6 | 4 | 10
  Gender: Non-binary | 0 | 0 | 1 | 1
  Gender: Did not answer | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 28 | 7 | 52
  Not Hispanic or Latino | 1 | 1 | 3 | 5
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 6 | 14 | 2 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 7 | 12 | 6 | 25
  More than one race | 1 | 3 | 2 | 6
  Unknown or Not Reported | 0 | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  Graduate/Professional | 4 | 7 | 1 | 12
  College | 12 | 16 | 4 | 32
  Some college | 1 | 1 | 2 | 4
  Associate degree | 0 | 0 | 0 | 0
  High school | 0 | 4 | 2 | 6
  Did not answer | 1 | 2 | 2 | 5
The Anxiety and Related Disorders Interview Schedule for DSM-5 (adult) Clinical Severity Rating [Mean (Standard Deviation); unit: units on a scale] — Clinical severity rating (CSR) of the primary diagnosis derived from the interview. CSR ratings range from 0 (absent) to 8 (very severely disturbing/disabling). The CSR takes into account intensity and frequency of the symptoms as well as interference of functioning.
  units on a scale | 5.1 (0.7) | 5.4 (0.8) | 5.0 (0.8) | 5.2 (0.8)
Hamilton Rating Scale for Anxiety (HAM-A) [Mean (Standard Deviation); unit: units on a scale] — The HAM-A is a clinician-administered 14-item measure of the severity of both psychic and somatic anxiety, with a total score range of 0-56. Total scores of ≤ 7 indicate no/minimal anxiety, 8-14 indicate mild anxiety, 15-23 indicate moderate anxiety, and ≥ 24 indicate severe anxiety.
  units on a scale | 14.3 (5.8) | 16.7 (7.3) | 11.5 (3.4) | 15.0 (6.5)
Hamilton Depression Rating Scale (HAM-D) [Mean (Standard Deviation); unit: units on a scale] — The 24-item HAM-D measures depressive symptoms and has a total score range of 0-76, with ≤ 7 indicating absence of depression, 8-14 indicating borderline to mild depression, 15-25 indicating moderate to marked depression, and ≥ 26 indicating severe to extreme depression.
  units on a scale | 15.9 (6.3) | 16.4 (6.2) | 14.4 (4.3) | 15.9 (5.9)
Anxiety Sensitivity Index (ASI) [Mean (Standard Deviation); unit: units on a scale] — The ASI consists of 18 self-report items across three domains (physiological, cognitive, and social concerns) assessing fear of the consequences of experiencing anxiety (anxiety sensitivity, or "fear of fear"). The toal score ranges from 0-72, with higher scores indicating greater anxiety sensitivity.
  units on a scale | 22.4 (13.3) | 28.1 (15.1) | 22.3 (12.4) | 25.3 (14.2)
Liebowitz Social Anxiety Scale (LSAS) [Mean (Standard Deviation); unit: units on a scale] — The LSAS is a 24-item self-report rating scale measuring social anxiety, with a total score range of 0-144. Lower scores indicate lower levels of social anxiety, and higher scores indicate higher levels of social anxiety.
  units on a scale | 47.1 (27.3) | 59.3 (26.8) | 44.2 (29.7) | 52.7 (27.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxious Symptoms From Baseline to End of Treatment (Week 6)
Description: Change in anxiety between the three incentive conditions will be measured using the Hamilton Rating Scale for Anxiety (HAM-A), a 14-item questionnaire measure of the severity of anxiety symptoms. The items measure both psychic anxiety and somatic anxiety, where higher scores, defined by a score range of 18-56, indicate a greater presence of symptoms and lower scores, defined by a score range of 0-17, indicate mild to no anxiety symptoms.
Time Frame: Baseline to week 6 (end of intervention)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Social Support | Gain Framed | Loss Framed
Number analyzed (Participants) | 18 | 30 | 11
units on a scale | 4.78 (1.03) | 6.93 (1.41) | 6.09 (1.54)

2. Primary Outcome: Change in Anxious Symptoms From Baseline to End of Treatment (Week 6)
Description: Change in anxiety between the three incentive conditions will be measured using the Anxiety Sensitivity Index (ASI). The ASI is an 18-item scale containing three subscales measuring physical, cognitive, and social concerns regarding anxiety. Higher scores, defined by a score range of 18-72, reflect greater self-reported concern and lower scores, defined by a score range of 0-17, reflect little self-reported concern.
Time Frame: Baseline to week 6 (end of intervention)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Social Support | Gain Framed | Loss Framed
Number analyzed (Participants) | 18 | 30 | 11
units on a scale | 7.22 (2.19) | 11.73 (2.16) | 12.27 (3.86)

3. Primary Outcome: Change in Anxious Symptoms From Baseline to End of Treatment (Week 6)
Description: Change in anxiety between the three incentive conditions will be measured using the the Leibowitz Social Anxiety Scale (LSAS). The LSAS is a 24-item scale measuring fear and avoidance across social situations with a total score range of 0-144. Higher scores, defined by a total score range of 50-95 or greater, indicate greater fear and avoidance severity and lower scores, defined by a total score range of 0-49, indicate mild to no fear or avoidance.
Time Frame: Baseline to week 6 (end of intervention)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Social Support | Gain Framed | Loss Framed
Number analyzed (Participants) | 18 | 30 | 11
units on a scale | 36.06 (5.72) | 43.77 (3.91) | 27.45 (7.14)

4. Secondary Outcome: Mean Number of Sessions Completed
Description: Mean number of sessions completed in the mobile app over the course of treatment. A greater number of sessions completed over the course of treatment will indicate greater engagement.
Time Frame: End of intervention (week 6)
Measure: Mean (Standard Error); unit: sessions
Arm/Group | Social Support | Gain Framed | Loss Framed
Number analyzed (Participants) | 18 | 30 | 11
sessions | 11.56 (0.20) | 10.67 (0.41) | 10.00 (0.88)

5. Secondary Outcome: Mean Rating Score on the Mobile Application Rating Scale
Description: The mean rating score is a average of four rating sub-scales (engagement, functionality, aesthetics, quality of information) on the uMARS throughout the intervention (average of week 1, 3, and 6) for each participant. The Mobile Application Rating Scale (uMARS) is a 26-item measure of mobile application engagement, functionality, aesthetics, quality of information, and perceived impact. The mean rating score has a total range of 1-5, with higher total scores, defined by a mean score of 4 or greater, indicating greater application feasibility and lower scores, defined by a mean score of 3 or lower, indicating poorer application feasibility.
Time Frame: End of intervention (week 6)
Population: 2 participants in the loss framed arm, and 1 participant in the gain framed arm had missing data from various timepoints for this measure, and therefore were not included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Social Support | Gain Framed | Loss Framed
Number analyzed (Participants) | 18 | 29 | 9
units on a scale | 4.19 (0.08) | 4.18 (0.10) | 3.91 (0.15)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Social Support | Gain Framed | Loss Framed
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/30 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/30 | 0/11
Other Adverse Events (participants affected / at risk) | 1/18 | 1/30 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Social Support (N=18) | Gain Framed (N=30) | Loss Framed (N=11)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
root canal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT05130281/Prot_SAP_000.pdf